CLINICAL TRIAL: NCT01581021
Title: Pedicle Screw Usage in Conventional Fixation Pattern Constructs Compared to Thoracic Hook Constructs in Adolescent Idiopathic Scoliosis Patients and Neuromuscular Ambulators
Brief Title: Pedicle Screw Usage in Conventional Fixation Pattern Constructs Compared to Thoracic Hook Constructs in Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Lawrence Haber, Chief Pediatric Orthopaedics/Associate Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-0110
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: randomized; controlled; hooks; screws
MeSH Terms: interventions — Pedicle Screws

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic Pedicle Screws (Active Comparator): Group treated with pedicle screws in the thoracic spine
  Interventions: Device: Pedicle screws
- Laminar Hooks (Active Comparator): Group treated with hooks in the thoracic spine
  Interventions: Device: Laminar Hooks

INTERVENTIONS:
Device: Pedicle screws — Screws that are placed into the pedicle of vertebral body.
  Arms: Thoracic Pedicle Screws
Device: Laminar Hooks — Hooks are placed over the lamina of the vertebral body
  Arms: Laminar Hooks

SUMMARY:
Scoliosis is a deformity in which there is an abnormal curvature of the spine. Surgery is the main method of correcting this deformity. Rods are attached to the spine to make it strait. There are two ways to fix these rods to the bone of the spine: laminar hooks or pedicle screws. Hooks are an older form of fixation and do not penetrate the bone, but are instead placed over a part of the vertebra called the lamina. Screws are newer and do penetrate the bone. Screws are placed into the part of the vertebra called the pedicle. Most surgeons think screws correct scoliosis better than hooks. The current literature agrees that screws are better for deformity correction in the lumbar spine and patients with severe deformity. There is disagreement in the literature regarding which works better in the thoracic spine in less severe deformity. There are no randomized, controlled trials in the literature that examine whether constructs that use hooks in the thoracic spine and screws in the lumbar spine (called hybrid constructs) work as well as all-screw constructs. This clinical study is a randomized controlled trial being conducted to evaluate treatment outcomes in patients with scoliosis undergoing surgical correction for their curves using either all-screw or hybrid constructs as fixation devices. The study population is limited to those with less severe deformity and the investigators' hypothesis is that hybrid constructs will be as acceptable as screws in terms of correction.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of adolescent idiopathic scoliosis or neuromuscular scoliosis
* Fusion to include six of more levels in thoracic, thoracolumbar, or lumbar region
* Less than 21 years of age
* Able to undergo surgery based on physical exam, medical history, and surgeon judgement
* Willing to comply with the follow-up clinical and radiographic evaluation schedules
* Informed consent signed by patient and parent or legal guardian

Exclusion Criteria:

* Scoliosis with curvature greater than 100 degrees or less than 40
* Smaller juvenile subjects weighing less than 30 kg
* Rigid curves
* Infection in the disc or spine, past or present
* Subject is pregnant
* Evidence of abuse of alcohol and/or illicit drugs
* Subject is prisoner
* Subject has evidence of tumor(s), malignant disease or other significant illness with decreased life expectancy
* Subject is immunocompromised or being treated with immunosuppressive agents

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2005-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence L Haber, MD, Principal Investigator — University of Mississippi Medical Center; Erika D Womack, BS MS, Study Director — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with adolescent idiopathic scoliosis were recruited at a University Mississippi Medical center clinic from Nov. 2005 to Dec. 2008.
Pre-assignment Details: After consent, the patient was given an identification number with the computer-generated randomized construct assignment. Enrolled participants might have been excluded from the study due to not being randomized.
Period: Overall Study
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks
Started | 29 | 29
Completed | 19 | 18
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 4 | 6
Not completed — More than 2 hooks in thoracic | 3 | 0
Not completed — Neuromuscular | 2 | 1
Not completed — Not Randomized | 1 | 2
Not completed — Lenke 6 Classification | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 27 | 55
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.62 (2.21) | 14.17 (2.21) | 13.90 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Main Thoracic Cobb
Description: X-rays measures the degree of curve in the thoracic spine.
Time Frame: 24 months post-operative
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks
Number analyzed (Participants) | 19 | 18
Degree
  Preoperative | 55 (6) | 58 (8)
  4 weeks post-operative | 15 (7) | 18 (8)
  24 months at final follow-up | 14 (6) | 23 (8)

2. Primary Outcome: Rotation
Description: The degree to which the spinal column is rotated from its normal position will be assessed.
Time Frame: 24 months post-operative
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks
Number analyzed (Participants) | 19 | 18
degree
  Preoperative | 15 (4) | 14 (4)
  24 month post-operative | 7 (3) | 11 (5)

3. Primary Outcome: Scoliosis Research Society-30 Survey
Description: Participants were administered a validated survey for evaluating patient quality of life and satisfaction with treatment. Total SRS-30 scores (max = 150) and the domains: function (max = 35), pain (max = 30), self-image (max = 45), mental health (max = 25), and satisfaction with management (max = 15) were analyzed on a scale from 1 (worst) to 5 (best). The mean was obtained by dividing maximum possible score by the number of questions answered.
Time Frame: 24 months post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks
Number analyzed (Participants) | 19 | 18
units on a scale
  Preoperative | 3.9 (0.2) | 3.9 (0.2)
  24 months post operative | 4.0 (0.2) | 4.1 (0.3)

4. Secondary Outcome: Mobilization and Pain Survey
Description: Using a numeric rating scale (0 = no pain and 10 = unbearable pain), patients were asked to estimate their experienced pain while at rest and when mobile by specifying a number on the scale.
Time Frame: 24 months post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks
Number analyzed (Participants) | 19 | 18
units on a scale
  Resting Pain Scale Preoperative | 2 (2.31) | 1.96 (2.49)
  Resting Pain Scale 24 mo Post-operative | 1.25 (1.86) | 1.0 (1.41)
  Mobilization Preoperative Pain Scale | 2.433 (2.74) | 2.16 (2.34)
  Mobilization 24 mo Postoperative Pain Scale | 1.25 (2.17) | 1.6 (1.55)

ADVERSE EVENTS:
Time Frame: No adverse events occurred.
Arm/Group | Thoracic Pedicle Screws | Laminar Hooks
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
The design of this study is a computer-generated randomized trial. Initially, the first 3 participants were not computer-randomized and therefore, these subjects had to be removed from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No